CLINICAL TRIAL: NCT06159829
Title: Determination of the Effect of Virtual Reality on Pain and Anxiety in Patients Undergoing Upper Endoscopy: A Randomized Controlled Trial
Brief Title: The Effect of Virtual Reality on Pain and Anxiety in Patients Undergoing Upper Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Figen EROL URSAVAŞ, Associate professor, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CankırıKUE
Record Dates: First submitted 2023-11-15; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Virtual Reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Virtual Reality glasses
  Interventions: Behavioral: experimental
- Control (No Intervention): Patients in the control group underwent upper endoscopy following the standard protocol.

INTERVENTIONS:
Behavioral: experimental — intervention group used VR with a natural landscape and relaxing musical accompaniment during the upper endoscopy procedure.
  Arms: Virtual Reality

SUMMARY:
Background: Virtual reality (VR) is a tool that uses three-dimensional computer graphics-based technologies to make an individual feel as if they are physically in the virtual environment by misleading their senses. In recent years, the use of VR has been widely used in clinical applications such as anxiety disorders, pain, and stress coping VR can be used to relieve acute pain and anxiety in hospitalized patients and was shown in several studies to reduce pain and anxiety levels Aim: to evaluate the effect of virtual reality on anxiety and pain in patients who underwent upper endoscopy without sedation.

Design: A single-centre, parallel-group, randomised control trial. Methods: The study sample consisted of 100 patients assigned to the intervention group (n=50) or control group (n=50) by stratified block randomization to control for sex distribution. During the upper endoscopy procedure, patients in the intervention group watched a video of natural scenery through virtual reality goggles. The study outcomes were anxiety and pain.

DETAILED DESCRIPTION:
Gastrointestinal (GI) diseases are an important public health problem in Turkey and worldwide.The prevalence of upper GI diseases in Turkey is reported to be 32.7%. A large-scale global study suggested that more than 40% of people have GI disease that affects quality of life and use of health services.

Although upper GI tract endoscopy is an important interventional procedure used in the diagnosis of diseases, it causes patients discomfort and anxiety. Different studies have indicated that 5.5%-48.3% of individuals undergoing upper GI tract endoscopy experience severe anxiety, 15.6%-51.6% experience moderate anxiety, and 78.9% experience mild anxiety. In addition, symptoms such as gagging, nausea, abdominal bloating, and pain can be seen during the endoscopy procedure. Anxiety and pain may affect a patient's compliance and tolerance of the procedure, resulting in the procedure being unnecessarily prolonged and potentially increasing the incidence of complications.

Intravenous sedative and analgesic agents are frequently used during endoscopic procedures. However, sedative agents may cause complications such as phlebitis, hypoxemia, airway obstruction, hypoventilation, hypotension, arrhythmia, and aspiration. Especially in short procedures such as upper GI tract endoscopy, sedation-free endoscopy was introduced both to prevent adverse effects and reduce costs. In addition, some patients do not want to receive sedation due to concerns such as loss of control, allergies, cardiac arrest, and inability to wake up. In such cases, non-pharmacological interventions can be used to increase the patient's comfort, compliance with the procedure, and tolerance in sedation-free upper endoscopies. One of these interventions is Virtual reality (VR). In recent years, the use of VR has been widely used in clinical applications such as anxiety disorders, pain, and stress coping.

The aim of our study was to evaluate the effect of VR on anxiety and pain in patients undergoing upper endoscopy without sedation. This study will help fill the literature gap and guide future research.

METHODS Trial design, participants and setting A single-centre, randomised controlled study was conducted in accordance with the CONSORT guideline. The population of the study comprised patients presenting to a city hospital in the Central Anatolia region of Turkey between June 22 and December 30, 2022 for upper endoscopy without anesthesia. The study sample consisted of 100 patients assigned to the intervention group (n=50) or control group (n=50) by stratified block randomization to control for sex distribution.

Sampling criteria

Patients meeting the following criteria were eligible for inclusion:

* Not using analgesics before the procedure,
* Not using anticoagulants within the last 24 hours,
* Having no vision or hearing problems
* Not receiving sedation
* Having no cognitive or psychiatric disorder that may affect understanding and communication Data collection Intervention Experimental protocol In addition to the standard protocol, patients in the intervention group used VR with a natural landscape and relaxing musical accompaniment during the upper endoscopy procedure. Before the procedure, the patients put on the VR goggles and started watching a video titled "4K Video Ultra HD - Breathtaking Sardinia" downloaded from youtube.com. They continued to watch the video throughout the endoscopy procedure, which lasted approximately 5 to 10 minutes. In both groups, levels of pain, state anxiety, and trait anxiety were measured and recorded before the procedure. After the procedure, the patients' pain levels and state anxiety levels during and after the procedure were assessed.

Standard protocol Patients in the control group underwent upper endoscopy following the standard protocol. In this protocol, written consent is obtained from the patient before the procedure and the patient is brought to the procedure room. The patient is asked about the use of anticoagulant agents, lidocaine spray is applied to the mouth to inhibit the gag reflex, and the mouthpiece is placed. The patient is placed in left lateral position for endoscopy, with left leg extended and right leg flexed towards the abdomen. The endoscopy procedure is then performed.

Data collection tools Data were collected using a sociodemographic and clinical information form, the Visual Analog Scale, and the State and Trait Anxiety Inventory.

Data analysis The data were analyzed using the free trial version of SPSS Statistics (Statistical Package for Social Sciences) for Windows version 25.0. Skewness and kurtosis values were examined to determine whether the data showed a normal distribution. The data were evaluated using descriptive statistics (number, percentage, mean, standard deviation) and compared between the groups using chi-square and independent-samples t tests.

ELIGIBILITY:
Inclusion Criteria:

* Not using analgesics before the procedure,
* Not using anticoagulants within the last 24 hours,
* Having no vision or hearing problems
* Not receiving sedation
* Having no cognitive or psychiatric disorder that may affect understanding and communication

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Comparison of mean pain scores of patients in the intervention and control groups of during endoscopy | Patients' pain levels were evaluated immediately after the procedure was completed.
  Visuel Analog Scale (VAS) This one-dimensional measure of pain intensity is a reliable and easily applicable scale that is widely accepted in the literature. VAS is used to convert nonmeasurable variables into numeric values. The 10cm scale is labeled 0 ("no pain") at one end and 10 ("extreme pain") at the other, with values indicated at each cm in between

SECONDARY OUTCOMES:
Comparison of mean anxiety scores of patients in the intervention and control groups of during endoscopy | Patients' anxiety levels were evaluated immediately after the procedure was completed.
  The anxiety inventory assesses how the person feels in certain circumstances and at a certain moment, while the trait anxiety inventory assesses how the person usually feels. Each item is scored between 1 and 4. A higher total score is interpreted as a higher level of anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Figen Erol Ursavaş, Principal Investigator — Cankırı Karatekin Univeristy
Locations (1):
- Figen Erol Ursavaş, Aksu, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No